CLINICAL TRIAL: NCT00408018
Title: An Open Label Multicentric Phase 1 Study of Selective Cyclin Dependent Kinase Inhibitor P276-00 in Patients With Advanced Refractory Neoplasms
Brief Title: Phase I Study of P276-00 in Patients With Advanced Refractory Neoplasms
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to terminate this study after 202 mg/m2 cohort was taken as MTD achieved in other study at 185 mg/m2
Sponsor: Piramal Enterprises Limited (Industry)
Responsible Party: Dr Himanshu Parikh, Piramal Life Sciences Limited
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P276-00/02/05
Record Dates: First submitted 2006-12-04; First posted 2006-12-05 (Estimated); Last update posted 2009-01-01 (Estimated); Status verified 2008-12

CONDITIONS: Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — P276-00

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: P276-00 — Potent Cyclin dependent kinase (cdk) cdk4 D1, cdk1 B and cdk9 T inhibitor

SUMMARY:
P276-00 is a molecule derived from Rohitukine, which through pre clinical assays was identified as a selective Cdk4-D1 and Cdk1-B inhibitor.The inhibition of these Cdks causes cell cycle arrest between the G1-S transition thus blocking the cell cycle events at an early stage of development. It therefore has the potential for being efficacious with lesser side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically and/ or cytologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective.
2. Patients of either sex, of all races and ethnic groups, and > 18 years of age.
3. ECOG (Eastern Cooperative Oncology Group) performance status ≤ 2 .
4. Patients with life expectancy of at least 4 months.
5. Patients must have normal organ and marrow function as defined below:

   * Hemoglobin ≥10 gm/dL
   * absolute neutrophil count ≥ 1,500/mL
   * platelets ≥ 100,000/mL
   * total bilirubin within normal institutional limits
   * AST/ALT ≤ 2.5 X institutional upper limit of normal (ULN)
   * creatinine within 1.5 times the upper normal institutional limits
6. The effects of P276-00 on the developing human foetus are unknown. For this reason women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of the study during the duration of study participation and for at least 4 weeks after withdrawal from the study.
7. Women who are nursing should not be included into the study
8. Concomitant medications for diabetes, hypertension, pain relief and any other co-existing conditions, except cancer, are permitted when the patient is on study medication. There should be no change in the dosage of these medications in the 2 weeks prior to day 1 of cycle 1, with the exception of dosages for pain relief medication. Changes in the dose of anti-emetics and diuretics may be made provided they will not interfere with probable adverse effects of investigational product.
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study (date of consent); or patients who have not recovered from adverse events (except grade 1 toxicities) due to agents administered more than 4 weeks earlier.
2. Patients having received any other investigational agents within 4 weeks prior to the date of consent and patients who have not recovered completely from the side effects of the earlier investigational agent.
3. Patients with known brain metastases should be excluded from this clinical trial.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to P276-00.
5. Patients having history of myocardial infarction or uncontrolled cardiac dysfunction during the previous 6 months.
6. Patients having diarrhea requiring anti-diarrheal therapy.
7. Patients having coagulopathy requiring anticoagulation.
8. Patients with uncontrolled but stable intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Women who are pregnant or nursing. P276-00 may have the potential for teratogenic or abortifacient effects. Since there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with P276-00, breastfeeding should be discontinued if the mother is to be treated with P276-00.
10. Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients are excluded from the study.
11. Patients requiring the use of concomitant medications that prolong the QT/QTc interval and/or are known to cause Torsades de Pointes (TdP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-03; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Safety assessment by Laboratory investigations (Hematology,Biochemistry, urinalysis), ECG, Holter monitoring,Physical examination | 2 years

SECONDARY OUTCOMES:
Tumor measurements,Pharmacokinetics, MALDI- TOF to study plasma peptide pattern | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Purvish M parikh, MD, DNB, PhD, Principal Investigator — Tata Memorial Hospital; Raghunadharao D, MD, DM, Principal Investigator — Nizam's Institute of Medical Sciences; Ravikumar Saxena, MD, Principal Investigator — Global Hospital
Locations (3):
- India (3):
  - Nizam's Institute of Medicai Sciences, Hyderabaad, Andhra Pradesh
  - Global Hospital, Hyderabad, Andhra Pradesh
  - Tata Memorial Hospital, Mumbai, Maharashtra